CLINICAL TRIAL: NCT00837161
Title: Pilot Study of MRI-Guided High Intensity Focused Ultrasound Ablation of Uterine Fibroids
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 994043
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Results first posted 2011-11-28 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Uterine Fibroids; Uterine Leiomyomata
Keywords: High Intensity Focused Ultrasound Ablation; Uterine Fibroids; Leiomyomata; Non-Invasive Treatment of Uterine Fibroids; MRI-Guided; Fibroids; Uterine Leiomyomata
MeSH Terms: conditions — Leiomyoma; Myofibroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Philips MR guided HIFU system (Experimental): Patient receiving HIFU treatment
  Interventions: Device: Philips MR guided HIFU system

INTERVENTIONS:
Device: Philips MR guided HIFU system — HIFU is the use of focused ultrasound energy to penetrate through soft tissue and causes localized high temperatures (55°C to 70°C) for a few seconds within the target producing well defined regions of protein denaturation, irreversible cell damage, and coagulative necrosis
  Other Names: Philips Sonalleve MR-HIFU system

SUMMARY:
Uterine fibroids (leiomyomas) are a common cause of heavy uterine bleeding and pain in reproductive aged women and are the most common cause of hysterectomy in the United States. Women are seeking new ways to treat symptomatic uterine fibroids that allow them to avoid surgery. This study is the first step in this quest. We will study the novel use of magnetic resonance imaging (MRI) in enhancing the safety of the FDA approved technique to treat fibroids called High Intensity Focused Ultrasound (HIFU). The term 'high intensity focused ultrasound' means using ultrasound to heat and to thermally destroy tissue, in this case, uterine fibroids. The MRI system will allow us to watch the ultrasound path during treatment and monitor the temperature increase in the fibroid tissue that comes during the procedure.

In this pilot study, women with symptomatic fibroids will undergo MRI guided HIFU and then have a hysterectomy. This will allow us to confirm studies done in animals which show that it is possible to destroy specific tissue without harming normal tissue surrounding the targeted area.

The purpose of this clinical study is to confirm the safety and treatment capabilities of the Philips MR guided HIFU system for ablation of uterine fibroids. This is a single arm pilot study of 10 women who will undergo hysterectomy after the HIFU procedure. This study design of hysterectomy after treatment has been requested by the FDA as part of IDE approval for this new device and mirrors what has been required for similar devices. Safety will be assessed by evaluating treatment accuracy, complications, and adverse events. Treatment capabilities will be assessed by evaluating the fibroid volume ablated and other factors related to the procedure feasibility and acceptance including procedure duration, time to return to normal activity, and pain scores at the time of the procedure.

Study population

The Philips MR-HIFU System is intended for ablation of uterine fibroid tissue in pre- or perimenopausal women with symptomatic uterine fibroids who desire a uterine-sparing procedure. Patients must have completed child bearing prior to enrolling in this study. Patients will be recruited by referral to gynecology and interventional radiology at the NIH Clinical Center. Candidates for enrollment will already have symptomatic uterine leiomyomas and be willing to undergo hysterectomy for treatment. It is estimated that of apparently eligible subjects, at least 30 women will have to be screened in person in order to identify 10 who will be eligible for this study. Other studies of fibroid treatments are currently ongoing at the NIH. Women who have been interested in, but have not been selected for enrollment in those studies and who appear to be eligible to this study will be contacted for potential enrollment.

Study design:

This study is a multi-center, single arm trial evaluating the safety and treatment capabilities of the Philips MR-guided HIFU system in the treatment of symptomatic uterine fibroid patients who are otherwise healthy women. All patients enrolled in the study will undergo hysterectomy within a window of 30 days following HIFU treatment. Patients who have symptomatic uterine fibroids, meet clinical indications for hysterectomy, are eligible according to the inclusion and exclusion criteria and provide informed consent will be enrolled in this study. This study design of treatment followed by hysterectomy has been requested by the FDA as part of IDE approval for this new device and mirrors what has been required for similar devices. It is anticipated that women will participate in the study for a 3 month period to include the screening, HIFU treatment, hysterectomy and post hysterectomy follow-up.

The methodology used for this HIFU device capitalizes on the thermal properties of volumetric ablation rather than point ablation used by other focused ultrasound systems. Thus it is anticipated that this device will have a shorter treatment time compared to other HIFU machines. This HIFU system, via real-time MR thermometry monitoring, has automated thermal feedback during the procedure which may enhance safety. This pilot study will not only assess the safety of this device but will enable us to delineate the treatment capabilities of this system for future use in patients who want uterine sparing non-surgical treatment for symptomatic fibroids.

DETAILED DESCRIPTION:
Uterine fibroids (leiomyomas) are a common cause of heavy uterine bleeding and pain in reproductive aged women and are the most common cause of hysterectomy in the United States. Women are seeking new ways to treat symptomatic uterine fibroids that allow them to avoid surgery. This study is the first step in this quest. We will study the novel use of magnetic resonance imaging (MRI) in enhancing the safety of the FDA approved technique to treat fibroids called High Intensity Focused Ultrasound (HIFU). The term high intensity focused ultrasound means using ultrasound to heat and to thermally destroy tissue, in this case, uterine fibroids. The MRI system will allow us to watch the ultrasound path during treatment and monitor the temperature increase in the fibroid tissue that comes during the procedure.

In this pilot study, women with symptomatic fibroids will undergo MRI guided HIFU and then have a hysterectomy. This will allow us to confirm studies done in animals which show that it is possible to destroy specific tissue without harming normal tissue surrounding the targeted area.

The purpose of this clinical study is to confirm the safety and treatment capabilities of the Philips MR guided HIFU system for ablation of uterine fibroids. This is a single arm pilot study of 10 women who will undergo hysterectomy after the HIFU procedure. This study design of hysterectomy after treatment has been requested by the FDA as part of IDE approval for this new device and mirrors what has been required for similar devices. Safety will be assessed by evaluating treatment accuracy, complications, and adverse events. Treatment capabilities will be assessed by evaluating the fibroid volume ablated and other factors related to the procedure feasibility and acceptance including procedure duration, time to return to normal activity, and pain scores at the time of the procedure.

Study population

The Philips MR-HIFU System is intended for ablation of uterine fibroid tissue in pre- or perimenopausal women with symptomatic uterine fibroids who desire a uterine-sparing procedure. Patients must have completed child bearing prior to enrolling in this study. Patients will be recruited by referral to gynecology and interventional radiology at the NIH Clinical Center. Candidates for enrollment will already have symptomatic uterine leiomyomas and be willing to undergo hysterectomy for treatment. It is estimated that of apparently eligible subjects, at least 30 women will have to be screened in person in order to identify 10 who will be eligible for this study. Other studies of fibroid treatments are currently ongoing at the NIH. Women who have been interested in, but have not been selected for enrollment in those studies and who appear to be eligible to this study will be contacted for potential enrollment.

Study design:

This study is a multi-center, single arm trial evaluating the safety and treatment capabilities of the Philips MR-guided HIFU system in the treatment of symptomatic uterine fibroid patients who are otherwise healthy women. All patients enrolled in the study will undergo hysterectomy within a window of 30 days following HIFU treatment. Patients who have symptomatic uterine fibroids, meet clinical indications for hysterectomy, are eligible according to the inclusion and exclusion criteria and provide informed consent will be enrolled in this study. This study design of treatment followed by hysterectomy has been requested by the FDA as part of IDE approval for this new device and mirrors what has been required for similar devices. It is anticipated that women will participate in the study for a 3 month period to include the screening, HIFU treatment, hysterectomy and post hysterectomy follow-up.

The methodology used for this HIFU device capitalizes on the thermal properties of volumetric ablation rather than point ablation used by other focused ultrasound systems. Thus it is anticipated that this device will have a shorter treatment time compared to other HIFU machines. This HIFU system, via real-time MR thermometry monitoring, has automated thermal feedback during the procedure which may enhance safety. This pilot study will not only assess the safety of this device but will enable us to delineate the treatment capabilities of this system for future use in patients who want uterine sparing non-surgical treatment for symptomatic fibroids.

Primary Outcome parameters:

1. Verifying with MR imaging that the location of the HIFU lesion matches the expected location (binary)
2. Verifying with MR imaging that no unintended lesions are formed as a result of the treatment (binary)
3. Examining the uterine capsule and surrounding areas for unintended damage during hysterectomy (binary)
4. Evaluating any complications or adverse events that result from the MR-guided HIFU treatment (categorical)
5. Comparing the actual MR-measured ablated volumes to MR thermal dose predicted volumes (categorical)
6. Comparing the ablated volumes from histology to MR thermal dose predicated volume (categorical)
7. Ensuring on histopathologic examination of the uterus that the zones treated by MR-guided HIFU treatment are indeed necrosed (binary)

Secondary Outcome Parameters:

1. Pain and discomfort scores immediately before, during and after HIFU treatment:
2. Length of Hospital Stay (LOS)
3. Return to Activity

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Recommended for Total Abdominal Hysterectomy
  2. Age between 18 and 59
  3. Weight less than 140kg (or 310lbs)
  4. Pre or peri menopausal with FSH less than 40 mIU/ml
  5. Uterine size less than 24 weeks based on MRI and physical exam assessment
  6. Symptom severity score greater than or equal to 50 by Spies Uterine Fibroid Questionnaire.
  7. Cervical cytology no more severe than low grade SIL
  8. History of uterine leiomyoma causing symptoms of bleeding, pressure, or pain, as defined by the ACOG practice bulletin (ACOG Practice Bulletin 1994):
  9. Dominant intramural fibroid greater than or equal to 3 cm and less than or equal to 16 cm on imaging.

EXCLUSION CRITERIA:

1. Other pelvic disease (mass indicated by history or MR imaging such as endometriosis, ovarian tumor, acute or chronic pelvic inflammatory disease)
2. Desire for future pregnancy
3. Significant systemic disease even if controlled
4. Pregnant or Positive pregnancy test
5. Hematocrit less than 25%
6. Extensive scarring along anterior lower abdominal wall (greater than 50% of area) or scar tissue or surgical clips in the direct path of the HIFU beam
7. MRI or MRI contrast agent contraindicated
8. Unable to quantify or measure fibroids on MR exam including nonenhancing fibroids
9. Fibroid or uterine calcifications
10. Dominant fibroid is pedunculated or greater than 5 cm submucosal
11. Communication barrier

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2009-01; Primary Completion 2010-02 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - St. Luke's Episcopal Hospital, Houston, Texas

REFERENCES:
- [Background] Fennessy FM, Tempany CM, McDannold NJ, So MJ, Hesley G, Gostout B, Kim HS, Holland GA, Sarti DA, Hynynen K, Jolesz FA, Stewart EA. Uterine leiomyomas: MR imaging-guided focused ultrasound surgery--results of different treatment protocols. Radiology. 2007 Jun;243(3):885-93. doi: 10.1148/radiol.2433060267. Epub 2007 Apr 19. PMID 17446521
- [Background] Flynn M, Jamison M, Datta S, Myers E. Health care resource use for uterine fibroid tumors in the United States. Am J Obstet Gynecol. 2006 Oct;195(4):955-64. doi: 10.1016/j.ajog.2006.02.020. Epub 2006 May 24. PMID 16723104
- [Background] Hindley J, Gedroyc WM, Regan L, Stewart E, Tempany C, Hynyen K, Mcdannold N, Inbar Y, Itzchak Y, Rabinovici J, Kim HS, Geschwind JF, Hesley G, Gostout B, Ehrenstein T, Hengst S, Sklair-Levy M, Shushan A, Jolesz F. MRI guidance of focused ultrasound therapy of uterine fibroids: early results. AJR Am J Roentgenol. 2004 Dec;183(6):1713-9. doi: 10.2214/ajr.183.6.01831713. PMID 15547216
- [Derived] Sri T, Steren AJ, Stratton P. Endometrial Cancer: Hidden Pathology in a Patient with Abnormal Uterine Bleeding and Known Leiomyoma. Gynecol Obstet Invest. 2015;80(4):272-5. doi: 10.1159/000370002. Epub 2015 Jan 27. PMID 25634727
- [Derived] Venkatesan AM, Partanen A, Pulanic TK, Dreher MR, Fischer J, Zurawin RK, Muthupillai R, Sokka S, Nieminen HJ, Sinaii N, Merino M, Wood BJ, Stratton P. Magnetic resonance imaging-guided volumetric ablation of symptomatic leiomyomata: correlation of imaging with histology. J Vasc Interv Radiol. 2012 Jun;23(6):786-794.e4. doi: 10.1016/j.jvir.2012.02.015. PMID 22626269
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/A_2009-CH-0063.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first High Intensity Focused Ultrasound (HIFU) treatment was on February 8, 2009 and the last patient was treated on March 5, 2010. 2 study sites enrolled patients, 2 from St. Lukes in Houston, TX and 9 from National Institutes of Health in Bethesda, MD.
Pre-assignment Details: Patients were screened prior to treatment and the primary exclusion criteria was either uterine size per gestational age or fibroid size.
Groups:
- HIFU Treated: Women indicated for total abdominal hysterectomy underwent a single Magnetic Resonance guided-High Intensity Focused Ultrasound (MR-HIFU) session for uterine fibroid ablation prior to surgery. Subjects were followed up until the date of hysterectomy, or for 30 days if hysterectomy was declined.
Period: Overall Study
Arm/Group | HIFU Treated
Started | 11
Completed | 9
Not Completed | 2
Not completed — refused hysterectomy | 2

BASELINE CHARACTERISTICS:
Arm/Group | HIFU Treated
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 46.7 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Treatment-related Adverse Events (AE) Per Subject Resulting From HIFU Treatment of the Uterine Fibroids
Description: The number of treatment-related Adverse Events (AE) reported during the study, divided by the total number of treated subjects. This corresponds to the mean number of treatment-related Adverse Events per subject. Relatedness of an AE to the treatment was judged case-by-case by the investigator.
Time Frame: end of follow-up (date of hysterectomy, at latest day 30 after treatment)
Population: Safety was assessed per protocol; all 11 participants were evaluated for adverse events after HIFU treatment.
Measure: Mean (Full Range); unit: treatment-related AE/patient
Arm/Group | HIFU Treated
Number analyzed (Participants) | 11
treatment-related AE/patient | 1.3 (1.3) [0 to 3]

2. Secondary Outcome: HIFU Treatment Equals Location Per Hysterectomy
Description: Count the number of participants in which both of the following conditions are satisfied: the fibroid treated area as shown on MRI images during treatment is the same as displayed on fibroids from histology slices after hysterectomy, and no unintended lesions are visible in the uterus.
Time Frame: Day 0, Hysterectomy
Population: All participants who underwent hysterectomy following MR-HIFU treatment were included in this endpoint measure. Patients who refused hysterectomy were not included.
Measure: Number; unit: participants
Arm/Group | HIFU Treated
Number analyzed (Participants) | 9
participants | 9

3. Secondary Outcome: Length of Time to Return to Normal Activities
Description: Length of time to return to normal activity measured in number of days from HIFU treatment. Assessed by patient interviews during follow-up.
Time Frame: end of follow-up (date of hysterectomy, at latest day 30 after treatment)]
Population: per protocol
Measure: Mean (Full Range); unit: days
Arm/Group | HIFU Treated
Number analyzed (Participants) | 11
days | 1.4 [1 to 3]

4. Secondary Outcome: Numerical Range Scale (NRS) of Pain Level
Description: Pain Scores obtained by patient self-assessment on a 0-10 scale, with 0 corresponding to no pain and 10 corresponding to maximum pain.
Time Frame: Treatment Day: Baseline, Recovery, Discharge; Follow-up: 24 hours, 48 hours, 72 hours, 1 week, 2 weeks
Population: Subjects were included into analysis at a given time point if they had not received hysterectomy yet prior to that time point.
  Analysed subject numbers were:
  from baseline up to including 72 hours: 11 subjects (per protocol population); at 1 week: 6 subjects; at 2 weeks: 4 subjects;
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | HIFU Treated
Number analyzed (Participants) | 11
units on a scale
  Treatment Day: Baseline | 1.3 (1.7) [0 to 5]
  Treatment Day: Recovery | 2.6 [0 to 6]
  Treatment Day: Discharge | 1.4 [0 to 6]
  24 hours after treatment | 2.4 [0 to 6]
  48 hours after treatment | 1.5 [0 to 5]
  72 hours after treatment | 1.3 [0 to 4]
  1 week after treatment | 1.2 [0 to 3]
  2 weeks after treatment | 1.5 [0 to 3]

5. Secondary Outcome: Discomfort Level
Description: Patient's self-assessed discomfort level on a 4-point scale, with: 0 = no pain; 1 = mild; 2 = moderate; 3 = severe.
Time Frame: Treatment Day: Baseline, Recovery, Discharge; Follow-up: 24 hours, 48 hours, 72 hours, 1 week, 2 weeks
Population: as for outcome 4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | HIFU Treated
Number analyzed (Participants) | 11
units on a scale
  Treatment Day: Baseline | 0.7 [0 to 2]
  Treatment Day: Recovery | 0.8 [0 to 2]
  Treatment Day: Discharge | 0.5 [0 to 2]
  24 hours after treatment | 0.8 [0 to 2]
  48 hours after treatment | 0.6 [0 to 2]
  72 hours after treatment | 0.7 [0 to 2]
  1 week after treatment | 0.3 [0 to 1]
  2 weeks after treatment | 1.3 [0 to 3]

ADVERSE EVENTS:
Time Frame: Feb 9, 2009 through March 9, 2010
Description: Adverse events assessed by patient questionnaire.
  Only unexpected adverse events were reported in the "Other" Adverse Event Field.
  All adverse events were reported including those not related to treatment.
Arm/Group | HIFU Treatment
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 6/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIFU Treatment (N=11)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Neck pain caused by positioning during treatment
Pain at Rib Cage or Chest Level (Musculoskeletal and connective tissue disorders) | 2 (4) — Pain caused by positioning during treatment
Right leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) — pain possibly due to positioning during treatment
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Pain most likely due to positioning during treatment
Rectal Bleeding (Gastrointestinal disorders) | 1 (1) — Bleeding unlikely caused by treatment
Fatigue (Reproductive system and breast disorders) | 1 (1) — not related to treatment
Diarrhea (Gastrointestinal disorders) | 1 (1) — Unlikely related to procedure
Shin discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) — Definitely related
pain right buttock (Musculoskeletal and connective tissue disorders) | 1 (1) — possibly related to treatment
Pruritis (General disorders) | 1 (1) — Not related to treatment
Nausea (Gastrointestinal disorders) | 1 (1) — Not related to treatment
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) — probably related to treatment positioning
Right foot swelling (Musculoskeletal and connective tissue disorders) | 1 (1) — possibly related
Fever (General disorders) | 1 (1) — Caught a cold before treatment
Cold (General disorders) | 1 (1) — Caught a cold before treatment
Constipation (Gastrointestinal disorders) | 1 (1) — Not related
Sharp burning pain at abdomen (Injury, poisoning and procedural complications) | 1 (1) — possibly related to treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less